CLINICAL TRIAL: NCT06744881
Title: The Effectiveness and Safety of CAPA - IVM in Ovulatory Infertile Women: a Pilot Study
Brief Title: CAPA - IVM in Ovulatory Infertile Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/24/DD-BVMD
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Ovulatory Infertile Women
Keywords: CAPA-IVM

STUDY DESIGN:
Intervention Model Description: A pilot study (in blocks of 5 participants per cohort and 4 cohorts in total)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- To evaluate the effectiveness and safety of CAPA-IVM in ovulatory infertile women in relation to the (Experimental)
  Interventions: Procedure: CAPA-IVM

INTERVENTIONS:
Procedure: CAPA-IVM — On days 2-4 of the menstrual cycle, after patients have consented to CAPA-IVM, they will undergo oocyte aspiration anytime thereafter but no later than day 6 of the cycle. Pre-maturation will last for 24-30 hours. ICSI will be used for insemination. Freeze-only on day 3 or day 5 and frozen embryo transfer will be performed on the subsequent cycle using HRT protocol with a maximum of 2 embryos transfer

SUMMARY:
In vitro maturation (IVM) is an assisted reproductive technology (ART) using minimal or no ovarian stimulation. In IVM, immature oocytes at the germinal vesical (GV) or metaphase I (MI) stage retrieved from small antral follicles are cultured to reach metaphase II (MII) (ASRM, 2021).

Since the first successful IVM baby was reported, subsequent studies have been mostly focused on patients with polycystic ovary syndrome (PCOS) to reduce the risks associated with ovarian stimulation such as ovarian hyperstimulation syndrome (OHSS), thromboembolic complications and ovarian torsion (Cha et al., 1991; Chian et al., 2000). Numerous IVM protocols have been applied with or without FSH or hCG priming and using one step or two steps culture system to gain the optimum oocyte maturation rate, blastulation rate and live birth rate (Sanchez et al., 2019; De Vos et al., 2021).

A randomized controlled trial (RCT) conducted on women with high antral follicle count, including women with PCOS, indicated that CAPA-IVM was non-inferior to conventional IVF (Vuong et al., 2020). Studies also showed that the mental and motor development of children born after IVM was similar to that of those born after IVF and naturally conceived (Nguyen et al., 2022; Vuong et al., 2022). Additionally, IVM is considered an effective treatment for women with gonadotropin resistant ovary syndrome to have children with their own oocytes (Le et al., 2021). IVM is also a viable option for fertility preservation for women with cancer in need of urgent treatment and contraindicated to hormonal stimulation (Grynberg et al., 2022).

There is little evidence on the effectiveness of IVM on women without PCOS. Junk et al have compared the effectiveness of IVM between women with polycystic ovaries (PCO) and polycystic ovary syndrome (Junk and Yeap, 2012). Women with PCO had significantly lower oocytes collected than those with PCOS (p<0,001), maturation rate, blastocyst development rate, and clinical pregnancy rate were comparable between two groups (Junk and Yeap, 2012). Another study indicated the maturation rate after standard IVM of ovarian tissue-derived oocytes collected from cancer patients was 8-67% (Segers et al., 2020). A study conducted by Kirillova on ovarian cancer patients with normal to high ovarian reserve showed that CAPA-IVM resulted in a higher maturation rate in ovarian tissue oocytes compared to standard IVM (56% vs 36%, p=0.0045) (Kirillova et al., 2021).

Recently, IVF/ICSI has been indicated in almost all infertility patients without PCOS. A randomized controlled trial on non-PCOS women with high antral follicle counts revealed no significant differences between IVM and conventional IVF regarding the ongoing pregnancy rate, live birth rate and the incidence of pregnancy and perinatal complications (Vuong et al., 2020). IVM offers numerous advantages due to the concept of using mild or no stimulation. The risk of ovarian hyperstimulation syndrome is largely eliminated, the cost of treatment is notably reduced. IVM is also more convenient as it requires fewer patient visits, ultrasounds and blood tests (Ho and Vuong, 2023).

Therefore, this pilot study is to evaluate the effectiveness and safety of CAPA-IVM in ovulatory infertile women and evaluate its success rate in relation to their ovarian reserve.

DETAILED DESCRIPTION:
1. Screening for eligibility and randomization

   * This trial will be conducted at My Duc Hospital, Ho Chi Minh City, Viet Nam.
   * Eligibility screening will be performed on the first visit.
   * Patients meeting the inclusion criteria will be invited to participate in the study. Patients will be provided with study information and consent forms. The investigator will collect signed consent forms from all participants.
2. Oocyte retrieval:

   On days 2-4 of the menstrual cycle, after patients have consented to CAPA-IVM, they will undergo oocyte aspiration anytime thereafter but no later than day 6 of the cycle.

   Cycle programming with oral contraceptives or progestogens, nor ovarian stimulation with rFSH or hMG preparations nor the use GnRH analogues are allowed. The use of oral contraceptives will be considered from the second cohort of patients onwards in case the timing/scheduling of the oocyte retrieval needs to be optimized. No hCG or GnRH agonist preparations will be administered for triggering ovarian maturation prior to oocyte retrieval.
3. Capacitation in vitro maturation The follicular aspirates are collected and filtered through a cell strainer. After collection, COCs are washed and transferred to a four-well dish, containing CAPA medium. Following 24 hours of incubation in CAPA media, COCs complexes are cultured in IVM medium for 30 hours. Following IVM culture, oocytes are mechanically and enzymatically denuded from their cumulus layers under a stereomicroscope and oocyte maturation is assessed under the inverted microscope
4. Fertilization:

ICSI will be used to fertilize mature oocytes. Embryos will be cryopreserved at the cleavage-stage embryo (day 3) if the patient has less than 4 embryos. Patients with 4 or more embryos will be counseled on blastocyst culture (day 5) according to the IVFMD protocol. All viable embryos will be cryopreserved.

ELIGIBILITY:
Inclusion Criteria:

* Ageing from 18 to 37.
* Women without PCOS:

  * Having regular periods: >24 days and <35 days.
  * And not having clinical hyperandrogenism or biochemical hyperandrogenism.
  * And not presenting with peripheral distribution of polycystic ovaries on ultrasound.
  * Antral follicle count 15 ≤AFC ≤ 24 and Anti-Mullerian Hormone 2,1 ≤ AMH ≤ 5 ng/mL)
* Having indication for ART
* First ART cycle.
* No ovarian stimulation 3 months prior to study entry
* Agree to have all embryos frozen on day 3 or day 5.
* Agree to transfer no more than 02 cleavage-stage embryos or 01 blastocyst-stage embryo in a subsequent embryo transfer.
* Agree to participate in the study (Agree to undergo CAPA-IVM).

Exclusion Criteria:

* Donor oocyte cycles.
* Uterine abnormalities (adenomyosis, leiomyoma (≥5 cm), bicornuate uterus, intrauterine adhesion).
* Prior ovarian surgery.
* Surgically extracted sperm (by PESA, TESE or micro TESE).

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of metaphase II oocytes available after CAPA-IVM culture | 24-48 hours after eggs retrieved
  This will be analyzed according to the patient's ovarian reserve

SECONDARY OUTCOMES:
Number of patients aspirated without oocytes | OR day
  Count the number of patients aspirated without oocytes
Number of patients without mature oocytes after CAPA-IVM | OR day
  Count the number of patients without mature oocytes
Number of patients without embryos | OR day
  Count the number of patients without embryos
Oocyte maturation rate | 24-48 hours after eggs retrieval.
  The oocyte maturation rate is calculated by dividing the number of MII oocytes after CAPA-IVM by the number of cumulus-oocyte complex (COC) retrieved
Fertilization rate | ICSI day
  Number of fertilized oocytes divided by the number of ICSI oocytes
Number of fertilized oocytes | 16-18 hours after ICSI
  Count the number of 2PN oocytes at 16-18 hours after ICSI
Number of day-3 embryos | 64±2 hours after ICSI
  Count the number of day-3 embryos at 64±2 hours after ICSI
Day-3 embryo rate | 64±2 hours after ICSI
  Number of day-3 embryos divided by the number of fertilized oocytes
Number of good quality day-3 embryos | 64±2 hours after ICSI
  Count the number of day-3 embryos graded as grade 1 and grade 2.
Number of day-3 embryos frozen | 64±2 hours after ICSI
  Count the number of day-3 embryos frozen
Number of day-5/6 embryos | 114±2/140±2 after ICSI
  Count the number of day-5 embryos at 114±2/140±2 after ICSI
Day-5/6 embryo rate | 114±2/140±2 after ICSI
  Number of day-5/6 embryos divided by the number of fertilized oocytes
Number of good quality day-5/6 embryos | 114±2/140±2 after ICSI
  Count the number of day-5/6 embryos graded as grade 1 and grade 2
Number of day-5/6 embryos frozen | 114±2/140±2 after ICSI
  Count the number of day-5/6 embryos frozen

CONTACTS AND LOCATIONS:
Locations (1):
- IVFMD - MyDuc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No